CLINICAL TRIAL: NCT00075764
Title: Phase III Randomized Trial of Anastrozole Versus Anastrozole and Fulvestrant as First Line Therapy for Post Menopausal Women With Metastatic Breast Cancer
Brief Title: S0226 Anastrozole With or Without Fulvestrant as First-Line Therapy in Postmenopausal Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000349337; U10CA032102 (NIH); S0226 (Other: SWOG); CAN-NCIC-MAC7 (Other: NCIC-CTG)
Record Dates: First submitted 2004-01-09; First posted 2004-01-13 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Active Comparator): Patients receive oral anastrozole once daily on days 1-28.
  Interventions: Drug: anastrozole
- Arm II (Experimental): Patients receive oral anastrozole as in arm I. Patients also receive fulvestrant intramuscularly on days 1, 14, and 28 during course 1 and then on day 28 of the subsequent courses.
  Interventions: Drug: anastrozole; Drug: fulvestrant

INTERVENTIONS:
Drug: anastrozole — Given orally
Drug: fulvestrant — Given intramuscularly
  Arms: Arm II

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using drugs such as anastrozole and fulvestrant may fight breast cancer by blocking the use of estrogen. It is not yet known whether anastrozole is more effective with or without fulvestrant in treating breast cancer.

PURPOSE: This randomized phase III trial is studying giving anastrozole together with fulvestrant to see how well it works compared to anastrozole alone as first-line therapy in treating postmenopausal women with metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the time to tumor progression in postmenopausal women with metastatic breast cancer treated with anastrozole with or without fulvestrant as first-line therapy.
* Compare the clinical benefit (complete or partial response, confirmed or unconfirmed, or stable disease ≥ 24 weeks) and overall survival of patients treated with these regimens.
* Compare adverse events in patients treated with these regimens.
* Determine the prognostic significance of estrogen receptor positivity and HER2/neu status in patients treated with these regimens.
* Determine parameters of estrogen and clinical pharmacology and estrogen levels in patients treated with these regimens.
* Compare anastrozole plasma levels at 8, 16, and 24 weeks in patients treated with these regimens (closed as of 4/16/2009).
* Compare estradiol serum levels at 8, 16, and 24 weeks in patients treated with these regimens (closed as of 4/16/2009).

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to prior adjuvant tamoxifen therapy (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral anastrozole once daily on days 1-28.
* Arm II: Patients receive oral anastrozole as in arm I. Patients also receive fulvestrant intramuscularly on days 1, 14, and 28 during course 1 and then on day 28 of the subsequent courses.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed for up to 4 years.

PROJECTED ACCRUAL: A total of 690 patients (345 per treatment arm) will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer meeting 1 of the following criteria:

  * Metastatic disease (M1)
  * Multiple sites of new disease that is clinically obvious metastatic disease (e.g., multiple sites of new osseous disease)
* Measurable or nonmeasurable disease
* No known brain or CNS metastases
* Hormone receptor status:

  * Estrogen-receptor positive* AND/OR
  * Progesterone-receptor positive* NOTE: *Positivity defined as estrogen binding of > 10 fmol/mg cytosol protein by ligand binding assay or positive by immunohistochemistry

PATIENT CHARACTERISTICS:

Age

* Not specified

Sex

* Female

Menopausal status

* Postmenopausal, as defined by 1 of the following:

  * Prior bilateral oophorectomy
  * More than 12 months since last menstrual period with no prior hysterectomy
  * At least 55 years of age with prior hysterectomy
  * Under 55 years of age with a prior hysterectomy without oophorectomy and with estradiol and follicle-stimulating hormone levels consistent with menopause

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* No bleeding diathesis (e.g., disseminated intravascular coagulation or clotting factor deficiency)

Hepatic

* INR ≤ 1.6

Renal

* Not specified

Other

* HIV negative
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the cervix, or adequately treated stage I or II cancer currently in complete remission

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior immunotherapy for recurrent or metastatic disease

Chemotherapy

* No prior chemotherapy for recurrent or metastatic disease
* More than 12 months since prior adjuvant or neoadjuvant chemotherapy
* No concurrent chemotherapy for malignancy

Endocrine therapy

* Prior adjuvant hormonal therapy allowed
* At least 12 months since prior adjuvant luteinizing hormone-releasing hormone (LHRH) analogues

  * Menstrual periods must not have resumed since LHRH therapy
* More than 12 months since prior adjuvant or neoadjuvant aromatase inhibitors (e.g., anastrozole, letrozole, or exemestane)
* More than 12 months since prior fulvestrant
* No prior hormonal therapy for recurrent or metastatic disease
* No other concurrent hormonal therapy for malignancy
* No concurrent hormone replacement therapy

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No long-term anticoagulant therapy (except antiplatelet therapy)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 695 (Actual)
Dates: Start 2004-04; Primary Completion 2012-12 (Actual); Study Completion 2018-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rita S. Mehta, MD, Study Chair — Chao Family Comprehensive Cancer Center; Theodore A. Vandenberg, MD, Study Chair — London Health Sciences Centre
Locations (426):
- United States (418):
  - Regional Medical Center, Anniston, Alabama
  - Providence Cancer Center at Providence Hospital, Mobile, Alabama
  - Alaska Regional Hospital Cancer Center, Anchorage, Alaska
  - Providence Cancer Center, Anchorage, Alaska
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Highlands Oncology Group - Springdale, Bentonville, Arkansas
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Glendale Memorial Hospital Comprehensive Cancer Center, Glendale, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Tibotec Therapeutics - Division of Ortho Biotech Products, LP, Marysville, California
  - University of California Davis Cancer Center, Sacramento, California
  - San Francisco General Hospital Medical Center, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Tahoe Forest Cancer Center, Truckee, California
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Memorial Hospital Cancer Center - Colorado Springs, Colorado Springs, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - Shaw Regional Cancer Center, Edwards, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - Middlesex Hospital Cancer Center, Middletown, Connecticut
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Eugene M. and Christine E. Lynn Cancer Institute at Boca Raton Community Hospital - Main Campus, Boca Raton, Florida
  - North Broward Medical Center, Deerfield Beach, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - West Florida Cancer Institute at West Florida Hospital - Pensacola, Pensacola, Florida
  - Northeast Georgia Cancer Care, LLC - Medical Oncology, Athens, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Cancer Center - Medical Oncology, Rome, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - Portneuf Cancer Center at Portneuf Medical Center, Pocatello, Idaho
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - Resurrection Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Sherman Hospital, Elgin, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Provena St. Mary's Regional Cancer Center - Kankakee, Kankakee, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - Hematology Oncology Consultants - Naperville, Naperville, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Clarian Arnett Cancer Care, Lafayette, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Heartland Oncology and Hematology, Council Bluffs, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Pennington Cancer Center at Baton Rouge General, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - Central Maine Comprehensive Cancer Center at Central Maine Medical Center, Lewiston, Maine
  - York Hospital's Oncology Treatment Center, York Village, Maine
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Caritas St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Caritas Holy Family Hospital, Methuen, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Upper Michigan Cancer Center at Marquette General Hospital, Marquette, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - St. Luke's Hospital Cancer Care Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Keesler Air Force Base Medical Center, Keesler Air Force Base, Mississippi
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Independence Regional Health Center, Independence, Missouri
  - Freeman Cancer Institute at Freeman Health System, Joplin, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Midwest Hematology Oncology Group, Incorporated, St Louis, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - New Hampshire Oncology - Hematology, PA at Payson Center for Cancer Care, Concord, New Hampshire
  - Center for Cancer Care at Exeter Hospital, Exeter, New Hampshire
  - New Hampshire Oncology - Hematology, PA - Hooksett, Hooksett, New Hampshire
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Elliot Regional Cancer Center at Elliot Hospital, Manchester, New Hampshire
  - Monmouth Medical Center, Long Branch, New Jersey
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Capital Health Regional Cancer Center, Trenton, New Jersey
  - St. Francis Regional Cancer Center, Trenton, New Jersey
  - Lovelace Medical Center - Downtown, Albuquerque, New Mexico
  - Hematology Oncology Associates, PC, Albuquerque, New Mexico
  - Presbyterian Cancer Treatment Center at Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - St. Vincent Cancer Center at St. Vincent Regional Medical Center, Santa Fe, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Finger Lakes Hematology and Oncology, Clifton Springs, New York
  - Bassett Healthcare Regional Cancer Program at Mary Imogene Bassett Hospital, Cooperstown, New York
  - Adirondack Cancer Care - Glens Falls, Glens Falls, New York
  - Union State Bank Cancer Center at Nyack Hospital, Nyack, New York
  - Dyson Center for Cancer Care at Vassar Brothers Medical Center, Poughkeepsie, New York
  - Cancer Center of Poughkeepsie, Poughkeepsie, New York
  - Hudson Valley Oncology Associates, Poughkeepsie, New York
  - Highland Hospital of Rochester, Rochester, New York
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Hope A Women's Cancer Center, Asheville, North Carolina
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - FirstHealth Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Zimmer Cancer Center at New Hanover Regional Medical Center, Wilmington, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - Trinity CancerCare Center, Minot, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Cleveland Clinic Beachwood Family Health and Surgery Center, Beachwood, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Cleveland Clinic Cancer Center, Independence, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Tod Children's Hospital, Youngstown, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - St. Charles Medical Center - Bend, Bend, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Dubs Cancer Center at Rogue Valley Medical Center, Medford, Oregon
  - Providence Cancer Center at PMCC, Medford, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Kaiser Permanente Health Care - Portland, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - St. Luke's Cancer Network at St. Luke's Hospital, Bethlehem, Pennsylvania
  - Delaware County Regional Cancer Center at Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Oncology Hematology Associates of Northern Pennsylvania, PC at Hahne Regional Cancer Center, DuBois, Pennsylvania
  - Easton Regional Cancer Center at Easton Hospital, Easton, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Guthrie Cancer Center at Guthrie Clinic Sayre, Sayre, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Scranton, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Mabry Center for Cancer Care at Regional Medical Center, Orangeburg, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - University of Tennessee Cancer Institute - Memphis, Memphis, Tennessee
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Martha Jefferson Hospital Cancer Care Center, Charlottesville, Virginia
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Auburn Regional Center for Cancer Care, Auburn, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Columbia Basin Hematology, Kennewick, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center, Spokane, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - Madigan Army Medical Center - Tacoma, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - Community Comprehensive Cancer Center at Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Center for Cancer Treatment & Prevention at Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Vince Lombardi Cancer Center at Aurora Lakeland Medical Center - Elkhorn, Elkhorn, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Mercy Regional Cancer Center, Janesville, Wisconsin
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Medical Consultants, Limited, Milwaukee, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - All Saints Cancer Center at Wheaton Franciscan Healthcare, Racine, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic - Sheboygan, Sheboygan, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Clinic - Wausau Center, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Riverview UW Cancer Center at Riverview Hospital, Wisconsin Rapids, Wisconsin
- Canada (8):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Northeastern Ontario Regional Cancer Centre, Greater Sudbury, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Cancer Care Program at Thunder Bay Regional Health Sciences, Thunder Bay, Ontario
  - St. Michael's Hospital - Toronto, Toronto, Ontario
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan

REFERENCES:
- [Derived] Bergqvist M, Nordmark A, Williams A, Paoletti C, Barlow W, Cobain EF, Mehta RS, Gralow JR, Hortobagyi GN, Albain KS, Pusztai L, Sharma P, Godwin AK, Thompson AM, Hayes DF, Rae JM. Thymidine kinase activity levels in serum can identify HR+ metastatic breast cancer patients with a low risk of early progression (SWOG S0226). Biomarkers. 2023 May;28(3):313-322. doi: 10.1080/1354750X.2023.2168063. Epub 2023 Jan 29. PMID 36647745
- [Derived] Mehta RS, Barlow WE, Albain KS, Vandenberg TA, Dakhil SR, Tirumali NR, Lew DL, Hayes DF, Gralow JR, Linden HH, Livingston RB, Hortobagyi GN. Overall Survival with Fulvestrant plus Anastrozole in Metastatic Breast Cancer. N Engl J Med. 2019 Mar 28;380(13):1226-1234. doi: 10.1056/NEJMoa1811714. PMID 30917258
- [Derived] Unger JM, LeBlanc M, Blanke CD. The Effect of Positive SWOG Treatment Trials on Survival of Patients With Cancer in the US Population. JAMA Oncol. 2017 Oct 1;3(10):1345-1351. doi: 10.1001/jamaoncol.2017.0762. PMID 28586789
- [Derived] Mehta RS, Barlow WE, Albain KS, Vandenberg TA, Dakhil SR, Tirumali NR, Lew DL, Hayes DF, Gralow JR, Livingston RB, Hortobagyi GN. Combination anastrozole and fulvestrant in metastatic breast cancer. N Engl J Med. 2012 Aug 2;367(5):435-44. doi: 10.1056/NEJMoa1201622. PMID 22853014

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 707 Patients underwent randomization. 12 were excluded: 9 did not have metastatic disease, 1 had previous chemotherapy, 1 was estrogen-receptor and progesterone-receptor negative, 1 did not undergo chest imaging. In addition, 1 patient withdrew consent.
  694 patients were included in the analysis.
Groups:
- Arm I Anastrozole: Patients receive oral anastrozole once daily on days 1-28.
  anastrozole: Given orally
- Arm II Anastrozole and Fulvestrant: Patients receive oral anastrozole as in arm I. Patients also receive fulvestrant intramuscularly on days 1, 14, and 28 during course 1 and then on day 28 of the subsequent courses.
  anastrozole: Given orally
  fulvestrant: Given intramuscularly
Period: Overall Study
Arm/Group | Arm I Anastrozole | Arm II Anastrozole and Fulvestrant
Started | 345 | 349
Completed | 0 | 0
Not Completed | 345 | 349
Not completed — Adverse Event | 5 | 12
Not completed — Death | 4 | 8
Not completed — Withdrawal by Subject | 28 | 18
Not completed — Progression | 269 | 274
Not completed — Still on treatment | 8 | 15
Not completed — Delinquent | 4 | 2
Not completed — Not protocol specified | 27 | 19
Not completed — Under review | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I Anastrozole | Arm II Anastrozole and Fulvestrant | Total
Number analyzed (Participants) | 345 | 349 | 694
Age, Continuous [Median (Full Range); unit: years] | 65 [36 to 91] | 65 [27 to 92] | 65 [27 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 345 | 349 | 694
  Male | 0 | 0 | 0
Prior adjuvant tamoxifen [Number; unit: participants]
  Yes | 139 | 141 | 280
  No | 206 | 208 | 414
Prior adjuvant chemotherapy [Number; unit: participants]
  Yes | 103 | 129 | 232
  No | 242 | 220 | 462
Measurable disease [Number; unit: participants]
  Yes | 188 | 188 | 376
  No | 157 | 161 | 318
Disease site [Number; unit: participants]
  Bone only | 76 | 75 | 151
  Visceral | 167 | 181 | 348
  Nonvisceral | 102 | 93 | 195
Time between diagnosis of primary and metastatic disease [Number; unit: participants] — Population: Only patients with non missing value of time between diagnosis of primary and metastatic disease will be included.
  participants
    None: number analyzed (Participants) | 337 | 339 | 676
    None | 141 | 122 | 263
    3 mo to < 5 yr: number analyzed (Participants) | 337 | 339 | 676
    3 mo to < 5 yr | 40 | 47 | 87
    5 to < 10 yr: number analyzed (Participants) | 337 | 339 | 676
    5 to < 10 yr | 68 | 66 | 134
    >= 10 yr: number analyzed (Participants) | 337 | 339 | 676
    >= 10 yr | 88 | 104 | 192
HER2 status [Number; unit: participants] — HER2 denotes human epidermal growth factor receptor type 2. Population: Only patients with available HER2 status data will be included in the analysis.
  participants
    Positive: number analyzed (Participants) | 295 | 297 | 592
    Positive | 25 | 31 | 56
    Negative: number analyzed (Participants) | 295 | 297 | 592
    Negative | 270 | 266 | 536

OUTCOME MEASURES:

1. Primary Outcome: Time to Tumor Progression
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target measurable lesions over the smallest sum observed (over baseline if no decrease during therapy) using the same techniques as baseline. Unequivocal progression of non-measurable disease in the opinion of the treating physician. Appearance of any new lesion/site. Death due to disease without prior documentation of progression and without symptomatic deterioration. From date of randomization to time of first documentation of progression, symptomatic deterioration or death due to any cause. Patients last known to be alive and progression free are considered at last date of contact.
Time Frame: Every 4 weeks while on treatment. Then every 3 months until progression, then six months for two years then annually until four years or until death, which ever occurs first.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I Anastrozole | Arm II Anastrozole and Fulvestrant
Number analyzed (Participants) | 345 | 349
months | 13.5 [12.1 to 15.1] | 15.0 [13.2 to 18.4]
Statistical Analysis 1: Comparison: Arm I Anastrozole vs Arm II Anastrozole and Fulvestrant; Test type: Other; p = 0.007, Log Rank; Two-sided stratified log-rank test; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.68 to 0.94]

2. Secondary Outcome: Clinical Benefit (CR, PR, Confirmed or Unconfirmed, or Stable Disease >= 24 Weeks).
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable, Does not qualify for CR, PR, Progression or Symptomatic Deterioration. Clinical Benefit = CR + PR + Stable >= 24 weeks
Time Frame: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Arm I Anastrozole | Arm II Anastrozole and Fulvestrant
Number analyzed (Participants) | 345 | 349
percentage of participants | 70 | 73

3. Secondary Outcome: Overall Survival
Description: From date of randomization to date of death due to any cause. Patients last known to be alive are censored at last date of contact.
Time Frame: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I Anastrozole | Arm II Anastrozole and Fulvestrant
Number analyzed (Participants) | 345 | 349
months | 41.3 [37.2 to 45.0] | 47.7 [43.4 to 55.7]
Statistical Analysis 1: Comparison: Arm I Anastrozole vs Arm II Anastrozole and Fulvestrant; Test type: Other; p = 0.049, Log Rank; A log-rank test, stratified according to prior or no prior tamoxifen therapy; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.65 to 1.00]

4. Secondary Outcome: Number of Patients With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Adverse Events (AEs) are reported by CTCAE version 3.0 terminology. For each patient, worst grade of each event type is reported. Grade3 (Severe), Grade4 (Life-threatening), Grade 5 (Fatal)
Time Frame: Patients were assessed for adverse events after each cycle (1 cycle = 28 days) while on treatment.
Population: Eligible patients who had received the protocol treatments were included in the adverse event summaries. Any CTCAE 3.0 event of Grade 3 (serious), Grade 4 (life threatening) or Grade 5 (fatal) which were deemed to be related to protocol treatment are included.
Measure: Number; unit: Participants
Groups:
- Arm I Anastrozole: Patients receive oral anastrozole once daily on days 1-28
- Arm II Anastrozole and Fulvestrant: Patients receive oral anastrozole as in arm I. Patients also receive fulvestrant intramuscularly on days 1 , 14, and 28 during course 1 and then on day 28 of the subsequent courses.
Arm/Group | Arm I Anastrozole | Arm II Anastrozole and Fulvestrant
Number analyzed (Participants) | 337 | 348
Participants
  ALT, SGPT (serum glutamic pyruvic transaminase) | 1 | 1
  AST, SGOT | 3 | 1
  Albumin, serum-low (hypoalbuminemia) | 1 | 1
  Alkaline phosphatase | 1 | 0
  Anorexia | 0 | 1
  Bilirubin (hyperbilirubinemia) | 1 | 0
  CNS cerebrovascular ischemia | 0 | 2
  Calcium, serum-high (hypercalcemia) | 1 | 0
  Cataract | 1 | 1
  Confusion | 0 | 1
  Constipation | 1 | 1
  Dehydration | 1 | 1
  Diarrhea | 2 | 1
  Dizziness | 1 | 2
  Dyspnea (shortness of breath) | 1 | 1
  Edema: limb | 1 | 1
  Fatigue (asthenia, lethargy, malaise) | 7 | 9
  Febrile neutropenia | 1 | 0
  Fracture | 1 | 2
  Glucose, serum-high (hyperglycemia) | 1 | 2
  Hemoglobin | 1 | 3
  Hemolysis | 1 | 1
  Hot flashes/flushes | 2 | 7
  Hypertension | 2 | 1
  Inf w/normal ANC or Gr 1-2 neutrophils - Blood | 1 | 0
  Inf w/normal ANC or Gr 1-2 neutrophils - UTI | 1 | 1
  Infection with unknown ANC - Urinary tract NOS | 0 | 2
  Insomnia | 0 | 1
  Joint-effusion | 0 | 2
  Leukocytes (total WBC) | 0 | 1
  Lymphopenia | 3 | 3
  Memory impairment | 1 | 0
  Mood alteration - agitation | 0 | 1
  Mood alteration - anxiety | 1 | 0
  Mood alteration - depression | 0 | 3
  Mucositis/stomatitis (functional/symp) - Pharynx | 1 | 0
  Muscle weakness, not d/t neuropathy - body/general | 1 | 0
  Nausea | 3 | 1
  Neurology-Other (Specify) | 1 | 0
  Neuropathy: sensory | 1 | 0
  Neutrophils/granulocytes (ANC/AGC) | 0 | 2
  Pain - Abdomen NOS | 1 | 2
  Pain - Back | 5 | 7
  Pain - Bone | 1 | 1
  Pain - Breast | 1 | 0
  Pain - Buttock | 1 | 0
  Pain - Chest wall | 0 | 1
  Pain - Chest/thorax NOS | 1 | 1
  Pain - Extremity-limb | 0 | 3
  Pain - Head/headache | 1 | 0
  Pain - Joint | 5 | 7
  Pain - Muscle | 3 | 0
  Pain - Neck | 0 | 1
  Pain - Pelvis | 0 | 3
  Pain-Other (Specify) | 2 | 1
  Platelets | 2 | 2
  Rash/desquamation | 1 | 1
  Sodium, serum-low (hyponatremia) | 0 | 1
  Speech impairment (e.g., dysphasia or aphasia) | 1 | 0
  Sudden death | 0 | 1
  Syncope (fainting) | 0 | 1
  Thrombosis/embolism (vascular access-related) | 3 | 1
  Thrombosis/thrombus/embolism | 6 | 7
  Tinnitus | 0 | 1
  Tumor flare | 0 | 2
  Urticaria (hives, welts, wheals) | 0 | 1
  Vomiting | 3 | 2
  Weight gain | 0 | 1

ADVERSE EVENTS:
Time Frame: Patients were assessed for adverse events after each cycle (1 cycle = 28 days) while on treatment.
Description: Eligible patients who had received the protocol treatments and who were evaluable for adverse event assessment were included in the adverse event summaries. Any CTCAE 3.0 event of Grade 3 (serious), Grade 4 (life threatening) or Grade 5 (fatal) which were deemed to be related to protocol treatment are included.
Groups:
- Anastrozole: Patients receive oral anastrozole once daily on days 1-28
- Anastrozole & Fulvestrant: Patients receive oral anastrozole as in arm I. Patients also receive fulvestrant intramuscularly on days 1 , 14, and 28 during course 1 and then on day 28 of the subsequent courses.
Arm/Group | Anastrozole | Anastrozole & Fulvestrant
Serious Adverse Events (participants affected / at risk) | 21/337 | 48/348
Other Adverse Events (participants affected / at risk) | 309/337 | 322/348
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anastrozole (N=337) | Anastrozole & Fulvestrant (N=348)
Blood/Bone Marrow-Other (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 2 | 1
Atrioventricular block - 2nd degree Mobitz Type II (Cardiac disorders) | 0 | 1
Cardiac-ischemia/infarction (Cardiac disorders) | 1 | 2
Left ventricular diastolic dysfunction (Cardiac disorders) | 0 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 0
Restrictive cardiomyopathy (Cardiac disorders) | 1 | 0
Dry eye syndrome (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 1
Ileus, GI (functional obstruction of bowel) (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 1
Obstruction, GI - Ileum (Gastrointestinal disorders) | 0 | 1
Obstruction, GI - Small bowel NOS (Gastrointestinal disorders) | 0 | 1
Pain - Abdomen NOS (Gastrointestinal disorders) | 0 | 2
Perforation, GI - Colon (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 1
Death not associated with CTCAE term - Death NOS (General disorders) | 1 | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 | 1
Pain - Chest/thorax NOS (General disorders) | 0 | 1
Pain-Other (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 2
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Blood (Infections and infestations) | 0 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Bone (Infections and infestations) | 0 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Lung (Infections and infestations) | 1 | 2
Inf w/normal ANC or Gr 1-2 neutrophils - Pleura (Infections and infestations) | 0 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - Skin (Infections and infestations) | 0 | 1
Inf w/normal ANC or Gr 1-2 neutrophils - UTI (Infections and infestations) | 0 | 3
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 0 | 1
Infection with unknown ANC - Rectum (Infections and infestations) | 0 | 1
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 0 | 3
Fracture (Injury, poisoning and procedural complications) | 0 | 5
Leukocytes (total WBC) (Investigations) | 1 | 0
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1 | 1
Platelets (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 2
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 6
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 0 | 4
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 | 2
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 | 2
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint-effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness, not d/t neuropathy - Extrem-lower (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain - Back (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain - Bone (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain - Joint (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain - Neck (Musculoskeletal and connective tissue disorders) | 0 | 2
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 4
CNS cerebrovascular ischemia (Nervous system disorders) | 0 | 1
Cognitive disturbance (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Hemorrhage, CNS (Nervous system disorders) | 1 | 0
Neurology-Other (Nervous system disorders) | 0 | 1
Somnolence/depressed level of consciousness (Nervous system disorders) | 0 | 2
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 0 | 1
Syncope (fainting) (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 1 | 1
Mood alteration - agitation (Psychiatric disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pain - Pleura (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 2
Thrombosis/thrombus/embolism (Vascular disorders) | 1 | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Anastrozole (N=337) | Anastrozole & Fulvestrant (N=348)
Hemoglobin (Blood and lymphatic system disorders) | 64 | 80
Constipation (Gastrointestinal disorders) | 89 | 110
Diarrhea (Gastrointestinal disorders) | 64 | 72
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 46 | 47
Heartburn/dyspepsia (Gastrointestinal disorders) | 26 | 15
Nausea (Gastrointestinal disorders) | 114 | 119
Pain - Abdomen NOS (Gastrointestinal disorders) | 41 | 47
Vomiting (Gastrointestinal disorders) | 60 | 57
Edema: limb (General disorders) | 72 | 89
Fatigue (asthenia, lethargy, malaise) (General disorders) | 203 | 220
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 26 | 21
Injection site reaction/extravasation changes (General disorders) | 4 | 48
Pain - Chest/thorax NOS (General disorders) | 27 | 52
Pain-Other (General disorders) | 83 | 108
Rigors/chills (General disorders) | 28 | 20
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 18 | 22
Infection-Other (Infections and infestations) | 40 | 47
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 36 | 25
AST, SGOT (Investigations) | 52 | 43
Alkaline phosphatase (Investigations) | 36 | 46
Creatinine (Investigations) | 36 | 47
Leukocytes (total WBC) (Investigations) | 37 | 34
Lymphopenia (Investigations) | 10 | 22
Platelets (Investigations) | 14 | 26
Weight gain (Investigations) | 31 | 42
Weight loss (Investigations) | 24 | 21
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 18 | 18
Anorexia (Metabolism and nutrition disorders) | 78 | 74
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 20 | 25
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 20 | 25
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 73 | 95
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 6 | 18
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 11 | 25
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 27 | 31
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 26 | 29
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 12 | 18
Pain - Back (Musculoskeletal and connective tissue disorders) | 135 | 130
Pain - Bone (Musculoskeletal and connective tissue disorders) | 93 | 113
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 35 | 47
Pain - Joint (Musculoskeletal and connective tissue disorders) | 152 | 153
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 80 | 79
Dizziness (Nervous system disorders) | 59 | 65
Neuropathy: motor (Nervous system disorders) | 27 | 21
Neuropathy: sensory (Nervous system disorders) | 69 | 92
Pain - Head/headache (Nervous system disorders) | 66 | 81
Confusion (Psychiatric disorders) | 19 | 15
Insomnia (Psychiatric disorders) | 95 | 97
Mood alteration - agitation (Psychiatric disorders) | 13 | 18
Mood alteration - anxiety (Psychiatric disorders) | 58 | 58
Mood alteration - depression (Psychiatric disorders) | 63 | 79
Urinary frequency/urgency (Renal and urinary disorders) | 8 | 20
Pain - Pelvis (Reproductive system and breast disorders) | 17 | 24
Vaginal dryness (Reproductive system and breast disorders) | 22 | 24
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 8 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 91 | 92
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 96 | 102
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 12 | 19
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 11 | 23
Pruritus/itching (Skin and subcutaneous tissue disorders) | 27 | 45
Rash/desquamation (Skin and subcutaneous tissue disorders) | 45 | 61
Sweating (diaphoresis) (Skin and subcutaneous tissue disorders) | 53 | 62
Hot flashes/flushes (Vascular disorders) | 154 | 189
Hypertension (Vascular disorders) | 49 | 53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes